CLINICAL TRIAL: NCT04708717
Title: Encoding Temporal Fine Structure for Cochlear Implants
Acronym: TFS4CIs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of Rochester (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Raymond Goldsworthy, Associate Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01DC018044 (NIH)
Record Dates: First submitted 2021-01-07; First posted 2021-01-14 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hearing Loss; Cochlear Implants
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation Rate (Experimental)
  Interventions: Behavioral: Stimulation Rate; Behavioral: Electrode Location
- Electrode Location (Active Comparator)
  Interventions: Behavioral: Stimulation Rate; Behavioral: Electrode Location

INTERVENTIONS:
Behavioral: Stimulation Rate — Psychophysical training listening to stimulation rate as a cue for auditory pitch perception. The intervention is the listening rehabilitative exercises. Exercises are completed daily as 30-minute sessions for 2 weeks.
Behavioral: Electrode Location — Psychophysical training listening to electrode location as a cue for auditory pitch perception. The intervention is the listening rehabilitative exercises. Exercises are completed daily as 30-minute sessions for 2 weeks.

SUMMARY:
The goal of this study is to improve music and speech perception for cochlear implant users. Presently, most cochlear implants discard the temporal fine structure of sound, which is information that is widely believed to contribute to both music and speech perception. The proposed work examines perceptual and physiological changes that occur once this information is provided to cochlear implant users in a clear and consistent manner.

DETAILED DESCRIPTION:
The study goal is to improve music and speech perception for cochlear implant users. The relevant health outcome is their quality of life. This proposal focuses on how well cochlear implant users can learn to use temporal fine structure if provided as a clear and consistent cue for music or voice pitch. Historically, cochlear implants have discarded temporal fine structure and have only transmitted timing information of relatively slow envelope fluctuations. Attempts have been made to restore temporal fine structure into cochlear implant stimulation, but it is unclear whether previous attempts were limited by implementation, lack of experience, or inherently by physiology. The proposed approach is unique in that it examines the perceptual and physiological plasticity that occurs when temporal fine structure is restored. Proposed research is organized into two aims, which examine the relative salience of stimulation place and rate for providing a sense of pitch (Aim 1) and the salience of dynamic-rate stimulation compared to conventional methods (Aim 2). Both aims combine perceptual learning, computer-controlled electrode psychophysics, electrophysiology, and computational neural modeling to characterize the plasticity of pitch perception in cochlear implant users.

Aim 1 examines the perceptual and physiological plasticity associated with place and rate of cochlear implant stimulation. Cochlear implant users hear an increasing pitch associated with increasing stimulation rate, but this effect is difficult to measure above 300 Hz. Most studies of psychophysical sensitivity to cochlear implant stimulation rate have not considered perceptual learning. Preliminary results show that the sense of pitch provided by stimulation rate improves with training. The proposed research examines perceptual sensitivity and physiological encoding throughout a crossover training study with training provided for pitch based on place and rate of stimulation. The primary hypothesis tested is that cochlear implant users have a latent ability to hear pitch associated with stimulation rate, but they require training to learn how to use this new information.

Aim 2 is to determine whether dynamic-rate stimulation provides better sensitivity and better physiological encoding of fundamental frequency compared to conventional stimulation methods based on amplitude modulation of constant-rate stimulation. In normal physiology, auditory-nerve activity phase locks to the temporal fine structure of sound. Since cochlear implants typically discard this information, it is unknown how well cochlear implant users can learn to use it if provided. Aim 2 focuses on the comparison between dynamic-rate stimulation in which stimulation rate is dynamically adjusted to convey temporal fine structure compared to conventional methods based on amplitude modulation of constant-rate stimulation. The primary hypothesis is that dynamic-rate stimulation provides better pitch sensitivity and better physiological encoding compared to amplitude modulation of constant-rate stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Cochlear implant users.

Exclusion Criteria:

* Younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Baseline electrode psychophysics prior to training. | Measure collected prior to training.
  Just-noticeable difference for pitch ranking based on stimulation cues. Pitch discrimination will be measured as provided independently by place and rate of cochlear implant stimulation, as well as in combination. Stimuli will be dual-electrode pulse trains, which probe place-pitch perception with greater resolution than possible with single-electrode stimulation. Two-alternative forced-choice procedures will be used in which participants judge which of two stimuli is higher in pitch. Frequency discrimination will be measured near condition frequencies of 110, 220, 440, 880, and 1760 Hz for each of the 4 stimulation conditions (place, rate, combined). Adaptive procedures will be used to measure 75% discrimination accuracy.
Midpoint electrode psychophysics. | Measure collected at 4-week midpoint during psychophysical training.
  Just-noticeable difference for pitch ranking based on stimulation cues. Pitch discrimination will be measured as provided independently by place and rate of cochlear implant stimulation, as well as in combination. Stimuli will be dual-electrode pulse trains, which probe place-pitch perception with greater resolution than possible with single-electrode stimulation. Two-alternative forced-choice procedures will be used in which participants judge which of two stimuli is higher in pitch. Frequency discrimination will be measured near condition frequencies of 110, 220, 440, 880, and 1760 Hz for each of the 4 stimulation conditions (place, rate, combined). Adaptive procedures will be used to measure 75% discrimination accuracy.
Endpoint electrode psychophysics. | Measure collected at 8-week endpoint following psychophysical training.
  Just-noticeable difference for pitch ranking based on stimulation cues. Pitch discrimination will be measured as provided independently by place and rate of cochlear implant stimulation, as well as in combination. Stimuli will be dual-electrode pulse trains, which probe place-pitch perception with greater resolution than possible with single-electrode stimulation. Two-alternative forced-choice procedures will be used in which participants judge which of two stimuli is higher in pitch. Frequency discrimination will be measured near condition frequencies of 110, 220, 440, 880, and 1760 Hz for each of the 4 stimulation conditions (place, rate, combined). Adaptive procedures will be used to measure 75% discrimination accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT04708717/Prot_SAP_000.pdf